CLINICAL TRIAL: NCT01573468
Title: A Randomized, Double-blind Study of Capecitabine Plus Tesetaxel Versus Capecitabine Plus Placebo as Second-line Therapy in Subjects With Gastric Cancer
Brief Title: Capecitabine/Tesetaxel Versus Capecitabine/Placebo as Second-line Therapy for Gastric Cancer
Acronym: TESEGAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOG301; 2010-022164-12 (EudraCT Number)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — tesetaxel; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine-tesetaxel (Experimental): 21-day cycle; tesetaxel 27 mg/m2 orally once on Day 1; capecitabine 1750 mg/m2/day orally in 2 equally divided doses on Days 1-14
  Interventions: Drug: Tesetaxel; Drug: Capecitabine
- Capecitabine-placebo (Active Comparator): 21-day cycle; placebo orally once on Day 1; capecitabine 1750 mg/m2/day orally in 2 equally divided doses on Days 1-14
  Interventions: Drug: Placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel 27 mg/m2 orally once on Day 1 of each cycle
  Arms: Capecitabine-tesetaxel
Drug: Placebo — Placebo orally once on Day 1 of each cycle
  Arms: Capecitabine-placebo
Drug: Capecitabine — Capecitabine 1750 mg/m2/day orally twice daily (in 2 equally divided doses) on Days 1-14 of each cycle
  Other Names: Xeloda

SUMMARY:
This study is being performed to evaluate the efficacy and safety of capecitabine in combination with tesetaxel versus capecitabine in combination with placebo as second-line treatment for patients with gastric cancer.

ELIGIBILITY:
Key inclusion criteria:

1. Histologically or cytologically confirmed gastric adenocarcinoma, including gastric or gastroesophageal-junction adenocarcinoma (Histologically confirmed adenocarcinoma of the lower esophagus acceptable with radiographic or endoscopic documentation of gastroesophageal-junction or proximal-stomach involvement.)
2. Measurable disease (revised RECIST) based on computed tomography, or nonmeasurable disease
3. ECOG performance status 0 or 1
4. Treatment with only 1 prior regimen (as first-line therapy) that must have included a fluoropyrimidine and a platinum-containing agent (Prior adjuvant or neo-adjuvant chemotherapy acceptable provided 6 months elapsed between the end of this therapy and the start of first-line therapy.)
5. Disease progression after the start of the 1 prior regimen based on computed tomography
6. Adequate bone marrow, hepatic, and renal function
7. Ability to swallow an oral solid-dosage form of medication

Key exclusion criteria:

1. Squamous cell gastric carcinoma
2. Bone-only metastatic disease
3. History or presence of brain metastasis or leptomeningeal disease
4. Operable gastric or gastroesophageal-junction cancer
5. HER2-positive disease if the patient has not previously been treated with an anti-HER2 agent
6. Uncontrolled diarrhea, nausea, or vomiting
7. Known malabsorptive disorder
8. Significant medical disease other than gastric cancer
9. Presence of neuropathy > Grade 1 (NCI Common Toxicity Criteria)
10. Prior treatment (including adjuvant therapy) with a taxane or other tubulin-targeted agent (indibulin, eribulin, etc.)
11. Prior radiation therapy to more than 25% of the bone marrow
12. Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway
13. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | When at least 508 events of death have occurred, which is estimated will occur 12 months after the date of randomization of the last patient

SECONDARY OUTCOMES:
Disease control rate | Estimated will be assessed 12 months after the date of randomization of the last patient
  The percentages of patients with complete or partial response of any duration or stable disease lasting at least 6 weeks from the date of randomization (revised RECIST)
Progression-free survival | Estimated will be assessed 12 months after the date of randomization of the last patient
  Calculated from the date of randomization to the date when disease progression is first documented or when the patient dies within 60 days of the last lesion assessment
Response rate in patients with measurable disease | Estimated will be assessed 12 months after the date of randomization of the last patient
  The percentages of patients with complete or partial response (revised RECIST)
Incidence of adverse events | Through 30 days after the last dose of study medication
  The percentages of patients who experience adverse events by specific adverse event term

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Krankenhaus Nordwest, Frankfurt, Germany
- National Cheng Kung University Hospital, Tainan, Taiwan